CLINICAL TRIAL: NCT00356837
Title: Diagnosing Extremity Fractures and/or Dislocations Using Ultrasound in Adult Patients Presenting to the Emergency Department
Brief Title: Diagnosing Extremity Fractures and/or Dislocations Using Ultrasound Presenting to the Emergency Department
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB terminated study due to non compliance with continuing review date.
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Responsible Party: John G. McManus, LTC,, USAISR
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-06-004
Record Dates: First submitted 2006-07-24; First posted 2006-07-26 (Estimated); Last update posted 2010-12-13 (Estimated); Status verified 2010-12

CONDITIONS: Fractures; Dislocations
MeSH Terms: conditions — Fractures, Bone; Joint Dislocations | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Those with extremity fractures.
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — use ultrasound to confirm diagnosis of extremity fractures

SUMMARY:
The purpose of this study is to determine the efficacy of ultrasound in diagnosing the presence or absence of extremity fractures or dislocations.

Hypothesis: Can ultrasound be used as an accurate and effective method for determining the presence or absence of extremity fractures or dislocations? Is there a difference in amount of pain experienced prior to and after the ultrasound?

DETAILED DESCRIPTION:
This prospective, multicenter cohort study. The sampling method will be a convenience sample of all adult patients presenting to the ED with symptoms concerning a fracture and/or dislocation of an extremity. Once a patient has been deemed an appropriate candidate for the study, written consent will be obtained from one of the Associate Investigators. Once consent has been obtained, a resident physician will perform the ultrasound examination on the affected extremity(s) and note their findings.

ELIGIBILITY:
Inclusion Criteria:

* clinical suspicion of a fracture and/or dislocation of an extremity
* Age Greater than 18 years
* English speaking
* able to give consent

Exclusion Criteria:

* Age less than 18 years, including emancipated minors
* Unstable patients with B/P below 90mmHg systolic
* Open, unstable, or suspected compound fracture
* Physician has reviewed X-Rays and made diagnosis before ultrasound could be done
* X-Rays will not be ordered
* Patient is pregnant
* Patient cannot give own consent
* English is not the patient's primary language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Estimated)
Dates: Start 2006-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Faster diagnosis and sooner definitive treatment for extremity fractures or dislocations. | 1 hour

SECONDARY OUTCOMES:
Unnecessary evacuation in the pre hospital combat setting. | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: John G. McManus, MD, Principal Investigator — US Army Institute of Surgical Research
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

REFERENCES:
- [Background] Kirkpatrick AW, Brown R, Diebel LN, Nicolaou S, Marshburn T, Dulchavsky SA. Rapid diagnosis of an ulnar fracture with portable hand-held ultrasound. Mil Med. 2003 Apr;168(4):312-3. PMID 12733676